CLINICAL TRIAL: NCT07189728
Title: The MagnaSafe-2 Registry: Assessing the Risks of Magnetic Resonance Imaging in Three Patient Groups: (1) an MRI at a Magnet Field Strength of 3-tesla, (2) a "Mixed-vendor" or a Same Vendor "Mixed-component" Platform at 1.5-tesla or 3-tesla, or (3) a System With an Abandoned, Epicardial, or Fractured Lead at 1.5-tesla.
Brief Title: The MagnaSafe-2 Registry: Assessing the Risks of Magnetic Resonance Imaging in Three Patient Groups
Status: Not yet recruiting | Type: Observational
Sponsor: The Scripps Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: Russo_MagnaSafe2
Record Dates: First submitted 2025-09-11; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Pacemakers; MRI Imaging; Implantable Cardioverter Defibrillator (ICD)
Keywords: pacemaker; MRI; implantable cardioverter defibrillator; abandoned cardiac leads; 3-tesla

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Diagnostic Test: MRI — The MagnaSafe-2 Registry is designed to determine the risks of MRI in patients with limited MRI access not previously addressed in peer-reviewed literature and to improve access for approximately 70% of whom are predicted to have a future clinical need for MRI.

SUMMARY:
SUMMARY OF THE CLINICAL PROTOCOL Background: The risks of Magnetic Resonance Imaging (MRI) at 1.5-tesla for patients with a non-MRI-conditional (NMRC) pacemaker have been documented, guidelines for clinical practice have been published by the Heart Rhythm Society, and the Medicare National Coverage Determination (NCD) has been modified to provide coverage for these patients (CAG-00399R4). However, for patients with an abandoned, epicardial, or fractured cardiac lead or subcutaneous array, with a "mixed-vendor" or same-vendor "mixed-component" CIED, or those undergoing MRI at 3.0-tesla with a device not labelled as MRI-conditional (MRC) for use at 3-tesla, the risks of MRI have not been determined.

Hypothesis: For patients with an MRC or NMRC pacemaker or defibrillator and specific indications or circumstances not presently addressed, the risks of MRI do not increase.

Purpose: The MagnaSafe-2 Registry is designed to determine the risks of MRI in patients with limited MRI access not previously addressed in peer-reviewed literature and to improve access for approximately 70% of whom are predicted to have a future clinical need for MRI.

Study Design: A prospective registry of patients undergoing clinically indicated MRI. The protocol is being developed in collaboration with the FDA's Center for Devices and Radiological Health, and an Investigational Device Exemption is being requested for event reporting and monitoring. Also, "Coverage with Evidence Development (CED)" has been requested from CMS.

Enrollment: Eligible patients are 18 years or older and have a MRC or NMRC pacemaker system from any manufacturer, (after 2001), with leads from any manufacturer (without date restriction), and if the ordering physician has determined that MRI is clinically indicated, the imaging method of choice, and NOT performed for the purpose of research. Exclusions are a leadless pacemaker, a device battery at "elective replacement indicator," or renal insufficiency (GFR <45 cc/min). All participants will be required to provide informed consent for the collection of data.

Methods: Patients will be enrolled in the registry at up to 30 clinical centers with: (1) an NMRC pacing system scheduled for MRI at a magnet field strength of 3-tesla, (2) an NMRC system due to a "mixed-vendor" or a same vendor "mixed-component" platform at 1.5-tesla or 3-tesla, or (3) an MRC or NMRC pacing system and an abandoned, epicardial, or fractured lead at 1.5-tesla.

Primary Endpoints: A new cardiac arrhythmia noted during the MRI scan, or a Troponin-T elevation (>upper limit of normal) at 18-24 hours post-MRI scan compared to baseline (obtained within 30 days before the MRI scan), Troponin-T levels pre-MRI. Secondary Endpoints: Death, generator or lead failure requiring immediate replacement, loss of pacing capture (pacing-dependent patients), partial or full generator-electrical reset, pacing lead threshold increase of ≥1.0 V, a P-wave amplitude decrease of ≥50%, an R-wave amplitude decrease of ≥50%, and a pacing lead impedance change of ≥50 ohms from baseline.

Sample Size: Using an event rate limit of ≤1%, 500 cases will be needed in each group to yield a 95% confidence interval of 0 to 1.0% if no events are observed. When a total of 500 cases have been enrolled in one group, enrollment in the other groups may be continued at the discretion of the investigators. The estimated study duration is 5 years, including enrollment and data analysis.

Clinical Implications and Impact: The anticipated results will support an amendment to the current HRS Expert Consensus Statement (2017) and Medicare NCD (April 2018) for the patient groups in the study.

DETAILED DESCRIPTION:
1. INTRODUCTION 1.1 Specific aims The specific aims of the MagnaSafe-2 registry are to document the risks of magnetic resonance imaging (MRI) at a scanner strength of 3-tesla for patients with a non-MRI-conditional (NMRC) pacing system, to document the risks of MRI at 1.5-tesla for patients with an abandoned lead, epicardial lead, fractured lead or subcutaneous array, and to document the risks of MRI at 1.5-tesla or 3-tesla for patients with a "mixed-vendor" or "mixed-component" Cardiovascular Implantable Electronic Devices (CIED) system. A "mixed-vendor" system is defined as a combination of leads and a generator, both labeled for use in the MRI environment but from different manufacturers, and as a result, considered NMRC. A "mixed-component" system is defined as leads and a generator from the same manufacturer but not labelled as MRC as a combined device.

The study is a prospective multicenter registry of patients undergoing clinically indicated MRI. We anticipate that the results of the MagnaSafe-2 registry will support a change in MRI access for the three patient groups that are not addressed in the current HRS Expert Consensus Statement on MRI in Patients with CIED (2017), and are not covered by the updated Centers for Medicare and Medicaid Services (CMS) National Coverage Determination (CAG-000399R-4; April 2018).

1.2 Background and Significance Overall, 3 million people in the United States have a cardiac pacemaker or an implanted defibrillator, with approximately 600,000 being implanted each year. While CIED placement has increased, MRI has also become the imaging modality of choice for the evaluation of an increasing number of diseases of the brain, spinal cord, heart, and musculoskeletal system. Previous investigators have estimated that after placement of a pacemaker or a defibrillator, a patient will have a 50-75% chance of requiring a clinically indicated MRI study.

MRI was once believed to pose a risk for patients with a CIED, including a pacemaker, an implantable cardioverter defibrillator (ICD), or a cardiac resynchronization device. Most safety concerns regarding MRI were focused upon the potential of radiofrequency (RF) induced thermal injury at the interface of a cardiac lead and the distal myocardial implantation site in the right atrium, right ventricle, or coronary sinus. As a result of these safety concerns, it was long recommended that patients with a CIED should not undergo MRI scanning, even when MR was determined to be the most appropriate imaging modality for a specific clinical problem or anatomic location. To provide optimal care to the increasing number of patients with a CIED, health care professionals must have the capability to perform an MRI with full knowledge of the possible risks of the examination and have appropriate access to imaging for CIED patients.

1.3 MRI in Patients with Cardiac Devices Over the past two decades, CIED generator-plus-lead systems have been developed by many manufacturers to limit the potential risks associated with MRI. Device-plus-lead systems with a low or acceptable theoretical risk to the patient when used under specific conditions are labeled MRC by the US Food and Drug Administration (FDA) Center for Devices and Radiological Health in response to a manufacturer's request, accompanied by corroborating safety data. In February 2011, the first MRC pacemaker and lead system (Medtronic Revo MRI SureScan with 5086 leads) was approved by the FDA for scanning at an MR field strength of 1.5-tesla. Since that time, more than 50 pacemakers and defibrillator systems have received MRC labelling by the FDA Center for Devices and Radiological Health for use in the MR environment, and guideline documents have been published by several cardiovascular and radiological professional societies worldwide to address care for CIED patients.

In 2017, two landmark studies addressing the risks of MRI for patients with NMRC pacemakers or defibrillators were published. In the MagnaSafe Registry, MRI was performed in 1000 cases in which patients had a pacemaker and in 500 cases in which patients had an ICD. This study did not identify any deaths, lead failures, losses of capture, or ventricular arrhythmias during an MRI. One ICD generator could not be interrogated after MRI and required immediate replacement; the device had not been appropriately programmed per protocol before the MRI. Six cases of self-terminating atrial fibrillation or flutter and six cases of partial electrical reset were noted, most with an established history of arrhythmia. Changes in lead impedance, pacing threshold, battery voltage, and P-wave and R-wave amplitude exceeded pre-specified thresholds in a small number of cases. Multiple MRI scans were not associated with an increase in adverse clinical events.

Nazarian and colleagues found that in 1509 patients with a CIED, no long-term clinically significant adverse events were reported after MRI. In nine MRI examinations (0.4%), the patient's device reset to a backup mode. The reset was transient in eight of the nine examinations. In one case, a pacemaker with less than 1 month left of battery life reset to ventricular inhibited pacing and could not be reprogrammed; the device was subsequently replaced. The most common notable change in device parameters (>50% change from baseline) immediately after MRI was a decrease in P-wave amplitude, which occurred in 1% of the patients. At long-term follow-up (results available for 63% of the patients), the most common notable changes from baseline were decreases in P-wave amplitude (in 4% of the patients), increases in atrial capture threshold (4%), increases in right ventricular capture threshold (4%), and increases in left ventricular capture threshold (3%). The observed changes in lead settings were not clinically significant.

In 2017, an expert consensus statement was published by the Heart Rhythm Society (HRS). The objective of this document was to provide "practical recommendations in appropriate detail for health care providers of various backgrounds for the management of patients with a CIED so that they could undergo imaging and treatments in a manner that balanced benefit and risk." This HRS consensus statement addressed the use of MRI for patients with an implanted MRC or NMRC pacemaker or defibrillator.

Inspired by the new HRS guidelines, the data from two large clinical registries, and the findings from several smaller studies, a formal request was made to CMS to revise the existing NCD regarding MRI for Medicare/CMS beneficiaries with a NMRC cardiac pacemaker or defibrillator, and to remove the "Coverage with Evidence Development" (CED) requirement. In response, the CMS Coverage and Analysis Group proposed that any MRI examination for patients with an implanted cardiac device that did not have FDA labeling specific for use in an MRI environment (or NMRC) would be covered only if the MRI field strength was less than or equal to 1.5-tesla, if it has been 6 weeks or more since device and lead implantation or any lead revision, if the patient was not pacing dependent, and if no fractured, epicardial, or abandoned leads were present.

After the submission of a subsequent rebuttal letter by an expert group in response to the proposed NCD changes, the CMS Coverage and Analysis group released a subsequent and final decision memorandum in April 2018. In that memorandum (CAG-00399R4), the covered MRI field strength for NMRC systems was changed to 1.5-tesla only, and the exclusion for both a minimum time from device and lead implantation to the time of MR scanning was dropped, as well as the exclusion for pacing-dependent patients. However, the exclusion for fractured, epicardial, and abandoned leads remained. In the NCD memorandum, the CMS group stated that there was insufficient data to comment on the safety of MRI with abandoned leads and that they would "continue to monitor peer-reviewed medical literature for further evidence development and can reconsider this exclusion when sufficient evidence emerges which allows for the reassessment of the benefits and harms." 1.4 Preliminary data

1.4.1 Imaging at 3.0-tesla: Recent studies have suggested that MRI at a field strength of 3.0-tesla may be performed with minimal or no risk if patients are appropriately screened before the scan, monitored during the scan, and if the device is reprogrammed pre-scan and post-scan according to established imaging protocols. Previously, five studies have reported the results of MRI at a field strength of 3-tesla in patients with a CIED not labelled for use at that field strength. A total of 362 MRI scans at a field strength of 3.0-tesla have been performed in 328 patients, with most scans focused upon imaging of the brain and spine. No study has reported a serious adverse event related to exposure to MRI at 3.0-tesla.

1. Naehle et al. performed 51 MRI scans of the brain at a field strength of 3-tesla in 44 patients and did not find an increase in post-scan troponin levels measured to identify myocardial thermal injury due to lead tip heating. In addition, no serious adverse cardiac events were reported. This study identified no clinically significant device setting changes, no new arrhythmias, or other adverse clinical events. The authors concluded that MRI access should not be withheld from patients with an NMRC CIED and with a clinical need for a 3.0-tesla MRI scanning.
2. Gimbel studied 14 patients who underwent 16 MRI scans at a field strength of 3.0-tesla. There were no restrictions for pacing-dependence or the anatomic region scanned. A programming strategy using a no-pacing mode in patients who were not pacing dependent, and asynchronous pacing at the highest output was used in pacing-dependent patients. Device interrogation was performed before the MRI, immediately after the MRI, and at 1-3 months after the MRI. For non-pacing-dependent patients, attempts were made to turn all device features off. In pacemaker-dependent patients, the device was programmed to asynchronous mode at the highest output for the duration of the scan to render the device resistant to exposure to MRI. The specific absorption rate (SAR) was limited to 2W/kg. In this study, no arrhythmias were noted, and no significant changes were noted in the device settings, pacing thresholds, sensing, or lead impedance.

1.4.2 MRI for patients with abandoned, fractured, and epicardial leads A recent review by Meier et al. summarized safety data for patients with a CIED and with an abandoned or epicardial lead who underwent clinically indicated MRI. The authors identified 21 publications reporting data from 656 patients with 854 abandoned and/or epicardial leads who underwent 929 MRI scans of various regions of the body and found no major adverse cardiac events. Two studies in this review measured troponin levels and did not identify a significant change in post-MRI-scan troponin levels. Studies on patients with fractured leads have also been conducted by Greenhill et al., who reported the results of 126 MRI scans at a field strength of 1.5-tesla in 80 patients, with 67 patients having abandoned leads and 13 having lead fragments. In this study, no adverse clinical events were reported.

Higgins et al performed a single-center retrospective study to examine the outcomes of patients who had a pacemaker or a defibrillator generator removed before MRI, thus rendering the pacing leads abandoned. Pacing threshold settings after generator reimplantation were later assessed, as well as clinical patient outcomes. A total of 19 patients underwent MRI after pacemaker generator removal with retained pacing leads. There was a mean of 1.63 abandoned leads at the time of imaging, and none of the leads were MRC. Most of the scans performed were of the central nervous system, including the brain and spine. There were no adverse events within 7 days of the MRI scan in any of the patients with an abandoned lead after device reimplantation. In addition, no lead malfunctions or clinically significant changes in pacing thresholds were noted.

2 INNOVATION 2.1 Study design

The proposed study, the MagnaSafe-2 Registry, is a prospective, multicenter registry designed to determine the risks of MRI in three groups of patients presently without access to clinically indicated MRI and not previously addressed in clinical investigations or peer-reviewed literature. The three groups of patients presently without adequate access to MRI are those with (1) a patient with CIED system scheduled for MRI at a magnet field strength of 3-tesla and labelled NMRC at that field strength, (2) a patient with an NMRC system due to a "mixed-vendor" or a same vendor "mixed-component" system scheduled for imaging at 1.5-tesla or 3-tesla, and (3) a patient with an MRC or NMRC pacing system and an abandoned lead, epicardial lead, fractured lead or subcutaneous array scheduled for clinically indicated MRI at a field strength of 1.5-tesla.

2.2 Enrollment Inclusion Criteria:

Patients will be included in the registry if they fulfill all the following criteria:

1. Age of 18 years or older
2. Able to provide informed consent for entry in the research registry
3. Have a CIED from any manufacturer implanted after 2001
4. Have cardiac leads from any manufacturer without an implant date limitation
5. Documentation that the patient's ordering physician has determined that an MRI at 1.5-tesla or 3.0-tesla of any anatomic region is clinically indicated without an acceptable alternative imaging technology
6. The patient is scheduled for that imaging procedure
7. MRI will be performed for clinical purposes, and not for the purpose of entry into this research protocol
8. In addition, groups within the protocol require that an enrolled patient will have:

   1. An NMRC CIED scheduled for MRI at 3.0-tesla with a CIED that is not MRC at that field strength.
   2. A "mixed-vendor" or same vendor "mixed-component" system that is NMRC because the generator and lead combination are not labeled as MRC for use in the MR-environment.
   3. A CIED and abandoned lead, a fractured cardiac lead, an epicardial lead, or a subcutaneous array.

2.3 Enrollment Exclusion Criteria:

Patients will not be included in the registry if they fulfill any of the following criteria:

1. A generator battery at the elective replacement indicator (ERI)
2. Renal insufficiency (GFR <45 cc/min)
3. In addition, all standard clinical exclusion criteria for MRI in patients without a cardiac device will be observed.
4. Standard clinical exclusion criteria include pregnancy, severe claustrophobia (not responsive to pre-procedure medications), morbid obesity (abdominal diameter of greater than 60 cm), and the presence of ferro-magnetic metallic objects (such as intra-orbital or intra-ocular retained metal fragments, and intracranial vascular clips and coils)

2.3.1 Conditions which do not require exclusion from the present protocol

1. Prior coronary stent placement (without minimum time from stent implant exclusion)
2. Prior non-coronary or peripheral vascular stent placement (including aortic stent grafts)
3. Vascular shunts
4. IVC filters for thromboembolic prophylaxis
5. Mechanical or bio-prosthetic heart valves, regardless of placement procedure
6. Prior coronary artery bypass grafting surgery (including associated sternal wires)
7. A retained temporary epicardial pacing wire after cardiac surgery
8. Prior joint replacement surgery
9. Left atrial appendage occlusion device placement
10. Atrial or ventricular septal defect closure device placement
11. Any other non-CIED MRC device 2.4 Group 1 - A patient with a CIED system not labelled for use at 3.0-tesla (NMRC) scheduled for MRI at a magnet field strength of 3.0-tesla

    1. Two landmark clinical studies previously addressed the risks of MRI for patients with an NMRC pacemaker or defibrillator at a magnet strength of 1.5-tesla. In these two studies, device or lead failure did not occur in any patient with an NMRC pacemaker or ICD who underwent clinically indicated MRI at 1.5-tesla, was appropriately screened and monitored, and had the device reprogrammed before the procedure following a prespecified protocol.
    2. Since that time, the number of 3.0-tesla MR scanners has increased significantly, and the clinical indications for MRI scanning at a field strength of 3.0-tesla have expanded as well.
    3. A 3.0-tesla MR scanner has increased image resolution when compared to a 1.5-tesla or lower field strength scanner, and 3.0-tesla imaging is presently preferred for several anatomical areas, including brain, spinal cord, heart, coronary stress perfusion, and some musculoskeletal indications.
    4. Some recently developed pacemakers and defibrillators are labelled as MRC by the US FDA for scanning at a scanner field strength of 3.0-tesla
    5. In the MagnaSafe-2 Registry, pre- and post-MRI device settings will be assessed in addition to Troponin-T levels at 18-24 hours post-MRI scan compared to baseline levels pre-MRI (obtained within 30 days before the MRI scan) and a measure of renal function (creatinine and calculated glomerular filtration rate (GFR), in addition to assessment of device settings pre- and post-MRI (pacing threshold, lead impedance, measured P-wave and R-wave voltage, and battery voltage).
    6. The results of the 3-tesla group of the MagnaSafe-2 Registry will allow for assessment of patient risk, myocardial thermal injury, and will facilitate a change in the Medicare NCD as well as a change in HRS guidelines and thus improve access to clinically indicated MRI at a magnet field strength of 3-tesla for these patients who require imaging.

2.5 Group 2 - Patients with an NMRC system due to a "mixed-vendor" or a same vendor "mixed-component" system scheduled for MRI at a scanner field strength 1.5-tesla or 3-tesla

1. It is proposed that for patients with an implanted pacemaker, cardioverter defibrillator, cardiac resynchronization therapy pacemaker, or cardiac resynchronization defibrillator with MRC FDA labeling at the time of product approval for use in an MRI environment, MRC imaging of any anatomic region may be performed if the cardiac device (known as the index device) is used in the MRI environment according to the product labeling or Indications for Use.
2. "Mixed-vendor" or a same vendor "mixed-component" results in a system being classified as NMRC, and as a result, a patient having limited access to clinically indicated MRI. It has been estimated that the proportion of mixed-vendor systems was 5.1% in 2022.
3. Previous studies have shown no clinically relevant changes in lead parameters between non-mixed and mixed generator lead combinations.
4. Small-scale studies showed no increased risks of adverse events in mixed systems compared to MRC systems.
5. In the MagnaSafe-2 Registry, the proposed study clinical endpoints will include an increase in Troponin-T levels at 18-24 hours post-MRI scan compared to baseline pre-MRI and a measure of renal function (creatinine and GFR) in this group, as well as new onset of atrial or ventricular arrhythmia.
6. The results of the "mixed-vendor" or "mixed-component" group of the MagnaSafe-2 Registry will allow for assessment of patient risk, myocardial thermal injury, and a change in HRS guidelines, and thus improved access to clinically indicated MRI for these patients.

2.6 Group 3 - Patients with an MRC or NMRC CIED and an abandoned cardiac lead, epicardial lead, fractured lead, or subcutaneous array scheduled for MRI at a magnet field strength of 1.5-tesla

1. Patients with an abandoned cardiac lead were excluded from previous studies assessing the risks associated with MRI in patients with pacemakers and defibrillators. The exclusion was not due to safety concerns, but rather the inability to interrogate the abandoned cardiac lead after MR scanning. Therefore, when CMS was asked to reconsider coverage in the updated NCD, the resulting and current decision memo (CAG-00399R4) excluded patients with an abandoned cardiac lead not due to safety concerns, but rather due to the paucity of available clinical outcome data.
2. Previous clinical investigations regarding cardiac device patients with abandoned cardiac leads undergoing MRI were limited to observation of clinical events alone, including a new onset of arrhythmia. However, myocardial stimulation resulting in arrhythmia represents only one concern. Lead heating resulting in myocardial thermal damage is another significant potential risk of MRI with an abandoned lead. The only method of assessing thermal injury to the myocardium is to obtain pre- and post-MR scan serum markers of myocardial injury, including Troponin-T values or an alternative marker of myocardial necrosis (such as Troponin-I).
3. In a recent meta-analysis, 656 cardiac device patients were studied, with 854 abandoned and/or epicardial leads who underwent 929 MRI scans of different anatomical regions; no scan-related major adverse cardiac events were documented (25). However, most patients in this analysis did not have a systematic determination of pre- and post-scan Troponin values.
4. In the MagnaSafe-2 Registry, the present proposed study, clinical endpoints will include Troponin-T levels at 18-24 hours post-MRI scan compared to baseline (obtained within 30 days before MRI) and a measure of renal function (creatinine and calculated GFR), as well as new onset of atrial or ventricular arrhythmia.
5. The results of the abandoned lead group of the MagnaSafe-2 Registry will allow for assessment of patient risk of arrhythmia and myocardial thermal injury. It is assumed that the resulting data will lead to a change in CMS guidelines within the current NCD, allowing for coverage and thus improved access to clinically indicated MRI for these patients.

3 APPROACH 3.1 Study overview: The MagnaSafe-2 Registry involves an MRI performed for clinical purposes at the discretion of the ordering physician and will follow a similar study design as the previously performed and reported MagnaSafe Registry. MRI for patients with an implanted cardiac device will only be performed when, in the opinion of the ordering physician, MRI is the imaging modality of choice without an acceptable alternative, and the decision to have the scan will not be part of this research protocol. Completion of the MagnaSafe-2 Registry inclusion/exclusion form by the ordering physician or qualified medical professional responsible for study enrollment will document that MRI has been requested as the clinically indicated diagnostic imaging modality of choice for a specific disease or anatomic region without acceptable alternative imaging technology. A patient with a CIED who is scheduled for a clinically indicated MRI will be invited to enroll in this research study if they fall into three clinical groups. Enrollment will be open to all eligible patients until the target enrollment of 500 patients has been reached in the "abandoned lead" group. After reaching target enrollment in Group 3 (epicardial leads, abandoned leads, subcutaneous array), enrollment will be limited to Group 2 (mixed vendor/component) and Group 1 (3.0-tesla imaging) if that group has not yet reached a maximum enrollment of 500 patients. In the MagnaSafe-2 Registry, up to 30 clinical sites will enroll patients. MRI-compatible equipment will be required to monitor vital signs (pulse oximeter and single-lead cardiac rhythm monitor) while performing MRI scans on patients with an implanted pacemaker. Recommendations from the HRS in 2017 will be incorporated into the performance of MRI where appropriate, and the coverage criteria of the 2018 CMS decision memo will be observed. This protocol is being developed in cooperation with the FDA Center for Devices and Radiological Health, and an IDE will be requested for event reporting/monitoring. Also, a change in the CMS/NCD has been requested for CED payment.

3.1 MRI protocol

1. A cardiologist, other qualified physician, or a qualified medical professional (such as a Nurse Practitioner, Physician's Assistant, or registered nurse) will review the medical record to determine suitability for study entry.
2. A signed written informed consent will be obtained.
3. The radiology technical staff will use standard screening procedures in use at the participating clinical site to evaluate the patient for non-research-related contraindications to MRI. These standard, non-research related contraindications include a cerebral aneurysm clip or coil, an infusion pump, neuro-stimulator, metal shavings in the eye, ferrous metal implants, transdermal drug patches with metallic backing, cochlear implants, an allergy to gadolinium, morbid obesity, pregnancy, and severe claustrophobia.
4. A qualified medical professional with advanced cardiac life support training, in addition to a non-MRI-safe "crash cart," will be available throughout the procedure to respond to an adverse clinical event; the emergency equipment will include a non-MRI-compatible defibrillator with transcutaneous pacemaker options; patients will be monitored throughout the procedure with continuous cardiac rhythm recording and transcutaneous pulse oximetry.
5. All patients will undergo device interrogation in the MRI suite, but outside of the magnet room (Zone II or III), immediately before the MRI scan, and again immediately following the MRI scan.
6. Results of the device interrogation will be collected by the staff at the performing center, recorded on an appropriate form, and the data will be transmitted to the coordinating center using a secure web-based data input system (REDCap/Scripps Research).
7. A copy of the device interrogation printouts or an electronic *.pdf document format will be uploaded to the secure web-based data input system.

3.3 Primary Endpoints A rise in Troponin-T at 18-24 hours post-MRI compared to baseline Troponin-T (obtained within 30 days before the MRI scan) in the absence of renal insufficiency (a GFR of <45ml/min), death, or generator or lead failure requiring immediate device replacement.

3.4 Secondary Endpoints: A new onset atrial or ventricular cardiac arrhythmia noted during the MRI scan, loss of pacing capture (for pacing-dependent patients), partial or full generator-electrical reset, pacing lead threshold increase of ≥1.0 V, a P-wave amplitude decrease of ≥50%, an R-wave amplitude decrease of ≥50%, a pacing lead impedance change (positive or negative) of ≥50 ohms from baseline, and patient reported heating, vibration, or discomfort at the generator implant site.

3.5 Sample Size Using a device failure or event rate of ≤1% as a limit, 500 cases will be needed in each group to yield a 95% confidence interval of 0 to 1.0% if no events are observed. When a total of 500 cases has been enrolled in one of the three groups, enrollment in the other 2 groups may be continued at the discretion of the investigators and the Data Safety Monitoring Board (DSMB).

3.6 Patient preparation Current clinical guidelines recommend removing and disposing of transdermal drug delivery patches before the MRI scan. As per standard individual institutional standards, all patients undergoing MRI must remove all readily removable metallic personal belongings, as well as clothing items which may contain metallic fasteners, hooks, zippers, loose metallic components, or metallic threads. The importance of having patients change into safe facility-provided garments before MR imaging is emphasized.

3.7 Examinations A case will be defined as an instance in which a patient who provides informed consent enters the scanner and undergoes an MRI of one or more anatomical regions during a single study session. If the patient returns on a subsequent day for a repeat MRI, then a separate informed consent will be obtained, and the data will be entered as a separate and unique case. No limit will be placed on the total number of repeat MRI examinations for an enrolled patient, the number of anatomic areas studied during each examination, or the interval between repeat MRI examinations during study enrollment. However, a patient may only be enrolled in one group of the study and may not return as part of a second or different study group.

3.7.1 Device programming during the scan:

1. The pacing rate will gradually be decreased to 40 bpm. If the patient has an intrinsic rhythm of greater than 50 bpm, then the patient will be determined to be not pacing-dependent, and the device will be programmed to a no-pacing mode (ODO or OVO).
2. If symptoms of lightheadedness or presyncope are noted, then the patient will be determined to pacing-dependent, and pacing function will be reprogrammed to an asynchronous pacing mode (DOO or VOO) at the previous baseline pacing rate or 60 bpm or greater.
3. If the patient has a generator which does not allow reprogramming to an ODO or OVO mode, and if the patient is not pacing-dependent, then the generator will be reprogrammed to an asynchronous pacing mode (DOO or VOO) and the pacing output for all active leads, and pulse-width should be set to a minimum value.
4. If there is an intrinsic rate of less than 50 bpm when the pacing rate is lowered to 40 bpm, then the patient will be determined to be pacing-dependent, and the device will be programmed to an asynchronous pacing mode (DOO or VOO) at the previous baseline pacing rate or 60 bpm or greater.
5. Patients with a cardiac resynchronization therapy pacemaker will be considered pacing-dependent regardless of the intrinsic rate and will be placed in an asynchronous pacing mode (DOO) at the baseline programmed rate for the duration of the MRI examination.

3.7.2 Pacemaker post-scan interrogation:

1. Post-scan generator interrogation will include a determination of the patient's underlying rhythm and a repeat interrogation of the device.
2. Post-scan interrogation of the device will include a measurement of the P and R wave amplitudes (if present at a pacing rate of 40 bpm) for all leads present; a measurement of the lead impedance for all leads (atrial, right ventricular, and left ventricular when present).
3. Pacing threshold measurements for all leads; pacing threshold measurements will be performed at 10 bpm above the programmed pacing rate or the patient's intrinsic rate. The pacing rate for testing can be increased by increments of 10 bpm if there is insufficient suppression of the patient's underlying rhythm.
4. Pacing threshold measurements will measure the pacing amplitude and will be performed with a fixed pulse width of 0.4 ms, regardless of the permanent pacing output. If the pulse width cannot be safely decreased to 0.4 ms to test a lead, the amplitude threshold test should be performed at the previously programmed or baseline pulse width.
5. Battery status will be interrogated after the scan, and the status (voltage or lifetime remaining) will be recorded.

3.7.3 Decision not to analyze battery status post-MRI scanning: When pre-MRI and post-MRI battery voltage measurements were compared in the first MagnaSafe Registry, a small decrease was noted for both pacemakers and ICDs. The RF energy generated during MRI scanning creates a temporary decrease in battery voltage, which has typically been reported to resolve within 2 weeks.

In the MagnaSafe Registry (2017), post-MRI battery voltage decreases of 0.04 V or more returned to baseline at the time of the last follow-up interrogation, which was typically between 3-6 months after the MRI scan. Thus, in the present study (MagnaSafe-2), the battery voltage, lifetime, or status will be measured and recorded post-MRI scan, but a change in battery voltage, lifetime, or status will not be used as a primary or secondary study endpoint.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included in the registry if they fulfill all the following criteria:

1. Age of 18 years or older
2. Able to provide informed consent for entry in the research registry
3. Have a CIED from any manufacturer implanted after 2001
4. Have cardiac leads from any manufacturer without an implant date limitation
5. Documentation that the patient's ordering physician has determined that an MRI at 1.5-tesla or 3.0-tesla of any anatomic region is clinically indicated without an acceptable alternative imaging technology
6. The patient is scheduled for that imaging procedure
7. MRI will be performed for clinical purposes, and not for the purpose of entry into this research protocol
8. In addition, groups within the protocol require that an enrolled patient will have:

   1. An NMRC CIED scheduled for MRI at 3.0-tesla with a CIED that is not MRC at that field strength.
   2. A "mixed-vendor" or same vendor "mixed-component" system that is NMRC because the generator and lead combination are not labeled as MRC for use in the MR-environment.
   3. A CIED and abandoned lead, a fractured cardiac lead, an epicardial lead, or a subcutaneous array.

      Exclusion Criteria:

      Patients will not be included in the registry if they fulfill any of the following criteria:

   <!-- -->

   1. A generator battery at the elective replacement indicator (ERI)
   2. Renal insufficiency (GFR <45 cc/min)
   3. In addition, all standard clinical exclusion criteria for MRI in patients without a cardiac device will be observed.
   4. Standard clinical exclusion criteria include pregnancy, severe claustrophobia (not responsive to pre-procedure medications), morbid obesity (abdominal diameter of greater than 60 cm), and the presence of ferro-magnetic metallic objects (such as intra-orbital or intra-ocular retained metal fragments, and intracranial vascular clips and coils)

      -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The proposed study, the MagnaSafe-2 Registry, is a prospective, multicenter registry designed to determine the risks of MRI in three groups of patients presently without access to clinically indicated MRI and not previously addressed in clinical investigations or peer-reviewed literature. The three groups of patients presently without adequate access to MRI are those with (1) a patient with CIED system scheduled for MRI at a magnet field strength of 3-tesla and labelled NMRC at that field strength, (2) a patient with an NMRC system due to a "mixed-vendor" or a same vendor "mixed-component" system scheduled for imaging at 1.5-tesla or 3-tesla, and (3) a patient with an MRC or NMRC pacing system and an abandoned lead, epicardial lead, fractured lead or subcutaneous array scheduled for clinically indicated MRI at a field strength of 1.5-tesla.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2031-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Troponin T levels | Baseline and 24 hours
  Troponin-T elevation (>upper limit of normal) at 18-24 hours post-MRI scan compared to baseline (obtained within 30 days before the MRI scan), Troponin-T levels pre-MRI.

SECONDARY OUTCOMES:
Arrythmia | Periprocedural
  Cardiac rhythm and oximetry will be monitored by qualified personnel (CV-MD, MD, PA, NP, or RN with pacemaker programming and ACLS training).
Changes to pacemaker | Periprocedural
  Measurement of battery voltage
Heart function | Periprocedural
  P-wave amplitude
Heart function | Periprocedural
  R-wave amplitude
Changes to pacemaker | Periprocedural
  lead impedance in ohms
Changes to pacemaker | Periprocedural
  pacing threshold settings for all leads in volts

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Russo, MD, PhD, Principal Investigator — Scripps Research

IPD SHARING:
Plan to Share IPD: Yes
The scientific data will be made available to other investigators upon appropriate request after the final database has been adjudicated and locked, and after first publication of the study results. The data will be stored and will remain available to appropriate investigators for 5 years following study publication.
  All patient data, including medical records, will be de-identified when possible, and unique study numbers will be used to refer to each patient enrolled in the study.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be stored and will remain available to appropriate investigators for 5 years following study publication following collection and locking of the database.
Access Criteria: Access to study data will be considered upon request to the coordinating center. NHLBI BioData Catalyst, a cloud-based system offering access in a secure workspace, will be utilized. Using this access portal, NHLBI-funded research/data may be reproduced by others to advance their scientific endeavors. When the results of the study are available, a manuscript will be submitted to the appropriate medical journal to achieve the best dissemination of the study results and conclusions. After the study, the results will be presented at either the annual scientific sessions of the American Heart Association and/or the American College of Cardiology. In addition, when the results of the study are available, results and conclusions will be posted at ClinicalTrial.gov.

REFERENCES:
- [Background] Russo RJ, Costa HS, Silva PD, Anderson JL, Arshad A, Biederman RW, Boyle NG, Frabizzio JV, Birgersdotter-Green U, Higgins SL, Lampert R, Machado CE, Martin ET, Rivard AL, Rubenstein JC, Schaerf RH, Schwartz JD, Shah DJ, Tomassoni GF, Tominaga GT, Tonkin AE, Uretsky S, Wolff SD. Assessing the Risks Associated with MRI in Patients with a Pacemaker or Defibrillator. N Engl J Med. 2017 Feb 23;376(8):755-764. doi: 10.1056/NEJMoa1603265. PMID 28225684
- See also: Lab website — https://www.ljcvri.org/